CLINICAL TRIAL: NCT00262652
Title: Sodium Pyruvate Bronchodilation in Asthmatics
Brief Title: Safety and Efficacy Study of the Use of Sodium Pyruvate Bronchodilation in Asthmatics
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patients did not respond to therapy
Sponsor: Emphycorp (Industry)
Responsible Party: Donald P. Tashkin, M.D., Professor of Medicine, David Geffen School of Medicine, UCLA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSI-UCLA-ASTHMA-01
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2005-11

CONDITIONS: Moderate Asthma
Keywords: sodium pyruvate; anti-inflammatory; bronchodilation; asthma; asthmatics
MeSH Terms: conditions — Asthma | interventions — BASS2 protein, Arabidopsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sodium pyruvate

SUMMARY:
Sodium pyruvate in sodium chloride solution will be delivered by nebulization to the lungs. It is believed that this administration will produce bronchodilation in asthmatics as determined by improvement in FEV1. FEV1 is a measure of lung function, and will be determined after administration of sodium pyruvate. The study is a blinded, so subjects may receive either the sodium pyruvate or a sodium chloride placebo. The primary endpoint will be the improvement of FEV1 after 15 minutes in subjects receiving sodium pyruvate compared to the FEV1 of subjects receiving the sodium chloride placebo.

DETAILED DESCRIPTION:
Sodium Pyruvate, an intermediate metabolite, has been investigated as a therapeutic agent to reduce reactive oxygen species in the lung. Evaluation of FEV1 as a safety parameter and sequela of reactive oxygen species reduction identified inhaled Sodium Pyruvate as a potential bronchodilator.

A number of lung diseases are typically characterized by marked inflammation at the site of the lung injury. This inflammatory process leads to further destruction of surrounding healthy lung tissue, and a continuation and expansion of the sites of inflammation. This inflammatory process results in the production of reactive oxygen species, including superoxide anions and hydrogen peroxide, at the site of inflammation.

Nitric oxide is a known bronchodilator, as well as a vasodilator. It has been used successfully used to treat patients with various pulmonary disorders. 1 When endogenous nitric oxide is exposed to oxygen radicals, however, it is converted to the toxic oxidant nitrogen dioxide, and its bronchodilating effect is mitigated. Conversely, nitrogen dioxide is a known deep lung irritant. Its adverse consequences include the following: pulmonary inflammation; reduced levels of lung antioxidants 2; impairment of respiratory defense mechanisms leading to increased susceptibility to respiratory pathogens 3 and increased incidence and severity of respiratory infections; reduced lung function, and increased asthma and COPD symptoms.

Reactive oxygen species, especially superoxide anions, are known to compromise lung function by increasing bronchoconstriction. As a result of the increasing inflammation and the production of reactive oxygen species, and the decrease in nitric oxide that is believed to occur with the interstitial lung diseases, healthy tissue is damaged and lung function is compromised.

Based on our present understanding of the disease process involved with these lung diseases, it appears that an intervention in the inflammatory process that would result in a reduction in reactive oxygen species and a subsequent increase in nitric oxide could be an effective way to intervene in the disease process. This intervention would prevent the further spread of inflammation and lung damage caused by the production of reactive oxygen species, such as superoxide anions and hydrogen peroxide, and increase lung function by increasing bronchodilation.

Sodium pyruvate is a reactive oxygen species antagonist that has been shown to neutralize oxygen radicals, specifically lowering the overproduction of superoxide anions, regulate the production and level of other inflammatory mediators, and increase the synthesis of nitric oxide. 4 Sodium pyruvate also increases cellular levels of glutathione, a major cellular antioxidant, which is reduced dramatically in antigen-induced lung disease patients. 5

In pilot studies in mild asthmatic subjects, it was demonstrated that inhalation of low doses (0.5 mM) of nebulized sodium pyruvate decreased expired hydrogen peroxide by 30% at four hours compared to inhalation of a nebulized saline control. These subjects also experienced increased pulmonary function as determined by FEV1 (+12.8%) and PEF (+34.5%) measurements after four hours (referenced in Cellular Sciences IND #50,089). It is theorized that the reactive oxygen species antagonist properties of sodium pyruvate reduced the production of oxygen radicals, including hydrogen peroxide, and increased the levels of nitric oxide. Together, this led to reduced inflammation and lung damage, and increased lung function through improved bronchodilation.

In summary, it is believed that inhalation of sodium pyruvate will reduce the lung damage resulting from the increase in reactive oxygen species associated with the inflammation component of the disease, and will enhances the availability of nitric oxide to produce bronchodilation by enhancing its synthesis and protecting it from destruction by reactive oxygen species.

Experimental Clinical Protocol Hypothesis: Sodium Pyruvate delivered by nebulization to the lungs produces bronchodilation in asthmatics as measured by FEV1

Intent: Provide support for further drug development of nebulized Sodium Pyruvate as a therapeutic agent in asthma

Design Randomized, double-blind, placebo-controlled cross-over study of 52 completed subjects

Treatment 1: 0.5 mM sodium pyruvate in 0.9% saline solution, (5ml) (Cellular Sciences, CA) nebulized via a Pari LC Plus(R) reusable nebulizer powered by a ProNeb(R) compressor (Midlothian, VA) Treatment 2: Saline 0.9%, (5ml) (Baxter) nebulized using the same nebulizer system as above A randomization algorithm using random permuted blocks (4-8 subjects) will be used to generate treatment order assignments. An unblinded statistician will generate this list of treatment order assignments.

Patient Recruitment and Selection The large cohort of potential subjects who have previously participated in asthma studies through our clinical research laboratory will be apprised of the study. Patients attending the UCLA Asthma and Cough Center will also be informed of the study. Advertisements will be sent by regular mail and by e-mail to physicians participating in the UCLA Healthcare System and to local pulmonologists practicing throughout the Los Angeles area. Local Allergists who collaborate with us in common clinical trial protocols will be informed of the study by personalized letter and e-mail. Advertisements will be placed in the classified and/or health sections of local newspapers. A description of the study will be posted on internet sites featuring clinical research trials.

Subjects will be recruited until a total of 52 complete the study. Assuming a 5% drop-out and non-compliance rate, we expect a total of 55 subjects recruited Patient Eligibility Criteria

ELIGIBILITY:
Inclusion Criteria:

1. A physician diagnosis of asthma
2. Age years old
3. Symptoms consistent with asthma for at least 6 months
4. Current asthma medications: Short-acting inhaled beta agonists as needed for control of asthma symptoms with or without a low to medium dose of an ICS, as defined in the table below and if on a ICS may also be on a long-acting beta agonist provided it is withheld for 24 hours prior to the testing days.

   Inhaled Corticosteroid Dose less than or equal to:

   Beclomethasone-HFA 480 µg/day Budesonide-DPI 1000 µg/day Flunisolide 2000 µg/day Fluticasone 500 µg/day Triamcinolone 2000 µg/day
5. FEV1 at screening 50-80% predicted (Hankinson6)
6. Reversibility with albuterol of 12% and 200 ml FEV1FEV1 at 30 minutes.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
ANCOVA using multiple measures evaluating FEV1% predicted at 5, 15, 30, 60, 120 and 240 minutes between saline and Sodium Pyruvate,and at 5, 15 and 30 minutes between albuterol and Sodium Pyruvate with the visit baseline FEV1% predicted as covariate. | Four Hour Testing
No other primary outcome variable

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tashkin, M.D., Principal Investigator — University of California, Los Angeles; Center for the Health Sciences
Locations (1):
- David Geffen School of Medicine, UCLA, Los Angeles, California, United States

REFERENCES:
- See also: Company Website — http://www.emphycorp.com/